CLINICAL TRIAL: NCT02955628
Title: A Phase II Study of Ibrutinib With R-ICE Chemotherapy for Transplant-eligible Relapsed/Refractory Diffuse Large B-cell Lymphoma Followed by Ibrutinib Maintenance in Patients Not Achieving a Complete Response at Pre-transplant Interim Assessment
Brief Title: RICE-ibrutinib in Relapsed DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGH-LYM-15-02
Record Dates: First submitted 2016-10-27; First posted 2016-11-04 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-11

CONDITIONS: Diffuse Large B Cell Lymphoma; Diffuse Large B-Cell Lymphoma Recurrent
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ibrutinib-RICE (Experimental): Patients not achieving a complete remission at time of PET-2 will receive ibrutinib and proceed on to autologous transplant if at least a partial remission is achieved. After transplantation, ibrutinib will be continued for up to 1 year. Autologous transplantation will be with BEAM conditioning.
  Interventions: Drug: Ibrutinib-RICE

INTERVENTIONS:
Drug: Ibrutinib-RICE — Ibrutinib will be added to RICE regimen for patients not achieving a complete remission at interim PET-2. Ibrutinib will be continued for up to 1 year after autologous transplantation.
  Other Names: Imbruvica

SUMMARY:
This is a multicentre, open-label, phase II study of ibrutinib 560 mg in combination with R-ICE for treatment of transplant-eligible relapsed/refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
All patients will receive R-ICE therapy for 2 cycles followed by PET-CT assessment (PET-2). Ibrutinib 560 mg will be added to the RICE regimen based on results of PET-2 as follows:

* Patients in CR will continue with 2 more cycles of R-ICE and proceed onto ASCT. These patients will not receive ibrutinib.
* In patients with stable disease or achieving a response that is less than CR, ibrutinib 560 mg will be added. The combination of ibrutinib-RICE will be given for 2 cycles and will be followed by PET-CT assessment (PET-4). Patients who achieve ≥ PR at this point will proceed onto ASCT.
* Patients who have disease progression will be removed from the trial. Hematopoietic stem cell harvesting can be performed following count recovery at any cycle of R-ICE, but preferably cycle 2.

Transplant conditioning regimen will be with standard BEAM chemotherapy (carmustine, etoposide, cytarabine, melphalan).

Following ASCT, ibrutinib will be given as maintenance therapy for patients who did not achieve a CR at the time of PET-2 assessment. This will be continued for up to 1 year after ASCT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven relapsed or refractory DLBCL (including transformed DLBCL)
2. Patients who are eligible for autologous stem cell transplant as deemed by the Bone Marrow Transplant Team in the participating cites.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (see Appendix A).
4. Minimum life expectancy of 6 months.
5. Previously treated with anthracycline-based chemotherapy (unless contraindicated) with rituximab Written informed consent
6. Must be at least 21 years old and able to sign informed consent form.
7. Adequate hematological function within 30 days prior to signing informed consent, including:
8. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L (1000/mm3) independent of growth factor support
9. Platelets ≥ 100,000/mm3 or ≥ 50,000/mm3 if bone marrow involvement independent of transfusion support in either situation
10. Hemoglobin ≥ 8 g/dL
11. Biochemical values within the following limits:
12. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN)
13. Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
14. Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockroft Gault) ≥ 40 mL/min/1.73m2
15. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
16. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
17. Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.
18. Must be able to adhere to study visit schedules and other protocol requirements.
19. Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

1. Concomitant use of any other investigational agent.
2. Contraindication to any drug contained in the regimen.
3. Myocardial infarction within 6 months prior to enrolment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
4. Clinically significant active infection.
5. Patients who are pregnant or breast-feeding.
6. Coexistent second malignancy or history of prior malignancy within previous 3 years (excluding non-melanoma skin tumors or in situ carcinoma of the cervix).
7. Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.
8. Major surgery within 4 weeks of randomization.
9. Known central nervous system lymphoma.
10. History of stroke or intracranial hemorrhage within 6 months prior to randomization.
11. Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon).
12. Requires treatment with strong CYP3A inhibitors.
13. Known inherited platelet function disorder.
14. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
15. Vaccinated with live, attenuated vaccines within 4 weeks of randomization.
16. Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
17. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by event free survival measured at 3-years follow up of patients who have received ibrutinib | 3 years
  Event-free survival is defined as time from diagnosis until relapse or progression, unplanned re-treatment of lymphoma after initial immunochemotherapy, or death as a result of any cause.

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival is defined as the time from enrolment to progression or death due to any cause. The distribution of PFS will be estimated using the method of Kaplan-Meier.
Overall survival | 3 years
  Overall survival is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Percentage of patients who have increased response from partial remission to complete remission ibrutinib before transplant | 6 weeks
  Reported as percentage of patients achieving a complete remission of the total patients starting ibrutinib.

CONTACTS AND LOCATIONS:
Locations (4):
- Singapore (4):
  - National University Hospital Singapore, Singapore
  - Singapore General Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
  - Raffles Hospital Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided